CLINICAL TRIAL: NCT03112122
Title: Randomized, Double-blind Study for the Treatment of the Bone Marrow Edema:Core Decompression Versus (VS) Subchondral Injections of Autologous BMC VS Subchondral Injections of Bone Substitute
Brief Title: Study for the Treatment of the Bone Marrow Edema:Core Decompression VS Bone Marrow Concentrate (BMC) VS Bone Substitute
Acronym: BME-TARGET
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Federica Balboni, Sub-Investigator, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BME-TARGET
Record Dates: First submitted 2017-03-30; First posted 2017-04-13 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Bone Marrow Edema
Keywords: Bone Marrow Edema; Mesenchymal Stem Cells

STUDY DESIGN:
Intervention Model Description: randomized, controlled, three-arm, double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- core decompression technique (Active Comparator): The standard surgical technique is the subchondral anterograde drilling, which permit a revascularization of the Bone Marrow Edema (BME) and a reduction of the intramedullary pressure (core decompression).
  Interventions: Procedure: core decompression
- bone substitution (i-FactorTM) (Experimental): i-FactorTM is a combination of the mineral component of bone (Anorganic Bone Mineral) with a peptide replicating the cell-binding domain of Type-I collagen (P-15). It has been used in bone defects and in spine fusion providing good clinical results. Thus, i-FactorTM could be a valid and efficient bone substitute to treat BMLs with subchondral injections.
  Interventions: Biological: bone substitute i-FactorTM
- injections of autologous Bone Marrow Concentrate (BMC) (Experimental): injections of autologous BMC.
  Interventions: Biological: autologous bone marrow concentrate

INTERVENTIONS:
Biological: autologous bone marrow concentrate — injection of autologous bone marrow concentrate
  Arms: injections of autologous Bone Marrow Concentrate (BMC)
Biological: bone substitute i-FactorTM — subchondral injections of i-FactorTM
  Arms: bone substitution (i-FactorTM)
Procedure: core decompression — subchondral anterograde drilling
  Arms: core decompression technique

SUMMARY:
Randomized, controlled, three-arm, double-blind study : control group, treated with core decompression technique VS subchondral plasty by injecting i-FactorTM VS injections of autologous BMC.

DETAILED DESCRIPTION:
The clinical trial is a randomized, controlled, three-arm, double-blind study, involving up to 120 patients. Eligible subjects will be randomly allocated to one of the three treatment groups: control group, treated with core decompression technique, study group 1, treated with subchondral plasty by injecting i-FactorTM, and study group 2, treated by injections of autologous BMC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18 and 75 years;
2. Symptomatic subchondral bone marrow lesions of femoral condyles (grade ≥ 1 according to the WORMS MRI score);
3. Failure after at least two months of a conservative treatment;
4. Single BME areas involving a single compartment of the knee;
5. Availability of the patients to participate actively in the rehabilitation protocol and follow-up clinic and radiology;
6. Signature of informed consent.

Exclusion Criteria:

1. Patients incapable of discernment;
2. History of allergy to calcium phosphates;
3. Patients with malignancies;
4. Patients with rheumatic diseases;
5. Patients with diabetes;
6. Patients suffering of metabolic disorders of the thyroid;
7. Patients with history of abuse of alcohol, drugs or medication;
8. Patients with advanced osteoarthritis (Kellgren-Lawrence grade> 3);
9. Body Mass Index> 35;
10. BME that involve more than one compartment;
11. Patients with trauma in the 6 months prior to the intervention. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
change of Visual Analogue Scale (VAS) score | [Timepoint: Screening, 1 , 3 6, 12, 24 months]
  improvement in VAS score from baseline to follow up

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) subjective score | [Timepoint: Screening, 1 , 3 6, 12, 24 months]
  improvement in IKDC subjective score from baseline to follow up
Knee Injury and Osteoarthritis Outcome (KOOS) Score | [Timepoint: Screening, 1 , 3 6, 12, 24 months]
  improvement in KOOS score from baseline to follow up
Tegner Activity Level Scale | [Timepoint: Screening, 1 , 3 6, 12, 24 months]
  improvement in activity level scale from baseline to follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No